CLINICAL TRIAL: NCT03981536
Title: A Multicenter, Open Label, Single-Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of AP-101 in Familial and Sporadic Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate AP-101 in Familial and Sporadic Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AL-S Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AP101-01
Record Dates: First submitted 2019-05-30; First posted 2019-06-11 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Familial Amyotrophic Lateral Sclerosis; Sporadic Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Amyotrophic lateral sclerosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AP-101: Dose Level 1 (Experimental): Single dose of AP-101
  Interventions: Drug: AP-101
- AP-101: Dose Level 2 (Experimental): Single dose of AP-101
  Interventions: Drug: AP-101
- AP-101: Dose Level 3 (Experimental): Single dose of AP-101
  Interventions: Drug: AP-101

INTERVENTIONS:
Drug: AP-101 — Administered by intravenous infusion (IV)

SUMMARY:
Single ascending doses of AP-101 will be administered by intravenous (IV) infusion

ELIGIBILITY:
Inclusion Criteria:

* All participants must adhere to contraception restrictions
* Female patients of non-childbearing potential due to:

  1. Menopause: spontaneous amenorrhea for at least 12 months not induced by a medical conditions such as anorexia nervosa and not taking medications that induced the amenorrhea (e.g., oral contraceptives, hormones, gonadotropin releasing hormones, anti-estrogens, selective estrogen receptor modulators, or chemotherapy)
  2. Surgical sterilization
* Have possible, probable, probable laboratory supported or definite and definite familial laboratory-supported ALS in accordance with the El-Escorial criteria
* Have familial or sporadic ALS.
* With onset of ALS symptoms, specifically onset of muscle weakness within past 48 months
* Have slow vital capacity (SVC) of (greater than or equal to) ≥60%
* If on riluzole, must be on a stable dose
* If on edaravone, must have completed 2 cycles and are expected to remain on the same dose throughout the study
* Able to provide informed consent. If the patient is not able to provide written consent due to aggravation of disease condition, written informed consent may be provided by a legally authorized representative
* Have venous access sufficient to allow for blood sampling
* Have clinical laboratory test results within normal reference range for the population or study site, or results with acceptable deviations that are judged to be not clinically significant

Exclusion Criteria:

* Are currently enrolled in, or discontinued from, within the last 30 days, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study
* Have a history or presence of medical illness including, but not limited to, any cognitive, cardiovascular, hepatic, hematological, renal, endocrine, or psychiatric, or any clinically significant laboratory abnormality that indicates a medical problem that would preclude study participation
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women who are lactating.
* Have undergone a tracheostomy unless it was removed at least 6 months prior
* Are on feeding tube, unless the insertion of a feeding tube is considered prophylactic
* Are on nasal intermittent positive pressure ventilation (NIPPV) >4 hours per day or at the discretion of the medical monitor
* Have undergone stem cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-11-02 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With One or More Non-Serious Adverse Events (AEs) or Any Serious AEs (SAEs) | Baseline up to day 84
  A clinical trial AE is any untoward medical event associated with the use of a drug or drug delivery system in humans, whether or not it is considered related to that drug or drug delivery system
Number of participants with abnormalities in vital signs, clinical laboratory assessments, physical or neurological examinations, or electrocardiograms (ECGs) | Baseline up to day 84
  Vital signs include blood pressure, pulse rate, and body temperature

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) | Baseline up to day 84
  In serum
Time of Maximum Drug Concentration (Tmax) | Baseline up to day 84
  In serum
Area Under the Concentration Time Curve (AUC) | Baseline up to day 84
  In serum
Pharmacokinetic Concentrations in Cerebrospinal Fluid (CSF) | Screening, and at either 1 hour, 4 hours, 24 hours, 48 hours, 72 hours, or 168 hours
  Taken at screening, and then only one sample per participant post-dose, in the higher level doses

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — AL-S Pharma SA
Locations (3):
- Canada (3):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Toronto, Ontario
  - Montreal Neurological Institute & Hospital, Montreal, Quebec